CLINICAL TRIAL: NCT00888472
Title: Safety and Efficacy of High-dose Leukocytapheresis Using a Large Filter in Patients With Refractory Asthma
Brief Title: Safety and Efficacy of High-dose Leukocytapheresis Using a Large Filter in Refractory Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gunma University (Other)
Responsible Party: Principal Investigator, Tamotsu Ishizuka, Clinical Professor, Gunma University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000001936
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Bronchial Asthma
Keywords: Extracorporeal leukocytapheresis
MeSH Terms: conditions — Asthma | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Leukocytapheresis

INTERVENTIONS:
Procedure: Leukocytapheresis — 5000 ml, the blood volume per body, treated once. Twice at an interval of 6 days.

SUMMARY:
Extracorporeal leukocytapheresis (LCAP) or granulocytapheresis (GCAP) has been used in the treatment of patients with rheumatoid arthritis and ulcerative colitis and has shown promising safety and efficacy. LCAP and GCAP seem to be effective for steroid-resistant inflammation. The investigators have already reported safety and efficacy of GCAP in refractory asthma and expect the beneficial effect of LCAP in refractory asthma. In this study, in order to improve the therapeutic effect of LCAP by increasing the quantity of leukocytes that were removed, the investigators conducted a clinical study to investigate safety and efficacy of high-dose LCAP performed using a larger filter and an increased dose of the blood volume per body weight treated, as an possible therapy for refractory asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilled the 2001 criteria for refractory asthma in American Thoracic Society.

Exclusion Criteria:

* Pregnant women.
* Patients with severe cardiovascular diseases.
* Patients with infective diseases.
* Patients with leukocytopenia or anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Improvement of morning peak flow rate (PEFR) or evening PEFR | 4 weeks after the treatment

SECONDARY OUTCOMES:
An improved score of asthma control test | 4 weeks after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tamotsu Ishizuka, M.D., Principal Investigator — Assistant Professor
Locations (1):
- Department Medicine and Molecular Science, Gunma University Graduate School of Medicine, Maebashi, Gunma, Japan